CLINICAL TRIAL: NCT00899301
Title: Breast Tissue/Body Fluids Repository
Brief Title: Collecting and Storing Tissue Samples From Women With or Without Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Professor of Radiation Oncology, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BRE 03103; P30CA068485 (NIH); VU-VICC-BRE-03103; VU-VICC-030747
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Breast Cancer
  Interventions: Other: biologic sample preservation procedure
- Patients without breast cancer
  Interventions: Other: biologic sample preservation procedure

INTERVENTIONS:
Other: biologic sample preservation procedure — Tissue, urine and blood collection.

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, blood, and urine from patients with or without breast cancer to study in the laboratory may help the study of cancer.

PURPOSE: This research study is collecting and storing tissue samples from women with or without breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To create a database that includes environmental, demographic, phenotypic, clinical, pathologic, genetic, and prognostic factors in large cohorts of women with different stages of breast cancer.
* To create a tissue repository that contains DNA, RNA, or protein from tumor tissue or normal tissue, peripheral blood lymphocytes, and plasma that are linked to frozen and/or paraffin-embedded pathology specimens.

OUTLINE: Patients undergo tumor tissue and normal tissue sample collection at the time of medically indicated surgery or biopsy. Archival tissue may also be collected. Patients and normal volunteers also undergo blood and urine sample collection. A repository of tissue, blood, and urine samples will be established to facilitate current and future research studies to learn about the biologic features of breast cancer development and progression. Research studies may include molecular pathology studies and gene and protein expression studies.

Patients' medical records are reviewed over approximately 5 years to determine if the test results are associated with health status. Patients do not receive the results of individual testing.

ELIGIBILITY:
* Breast lesion which is suspected to be cancer or a known diagnosis of breast cancer (any stage, at any point in the disease trajectory) who agrees to donate tissue/body fluids.
* Individuals of all races and ethnic groups are eligible for this trial. There is no restriction regarding age, race, or ethnicity. The trial is open to the accrual of men and women.
* Must sign informed consent for study of tumor specimens as part of a research project.
* Must give permission for their tumor specimens to be obtained from outside institutions for molecular analyses.
* Must be willing to be followed for recurrence, relapse and death from disease.

ELIGIBILITY CRITERIA FOR OPTIONAL PHYSICAL FUNCTION AND COGNITIVE ASSESSMENTS

* Must be 60 years of age or older
* Have completed initial round of cancer treatment
* Have completed the optional online survey and opted-in for the physical function and cognitive assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2004-01-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Creation of a tissue repository that contains DNA, RNA, or protein from tumor tissue or normal tissue, peripheral blood lymphocytes, and plasma that are linked to frozen and/or paraffin-embedded pathology specimens | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/